CLINICAL TRIAL: NCT06468631
Title: The Impact of Improving Clinical Patient Handover Interventions on Patient Outcomes and Handover Practices: A Complex Nursing Intervention Study
Brief Title: Effects of Nursing Patient Handover
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, SERAP GÜNGÖR, Lecturer, Kahramanmaras Sutcu Imam University
Other Study IDs: Handover
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Patient Satisfaction; Nurse's Role
Keywords: handover; handoff; patient safety
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Complex Nursing Intervention — Training prepared as an expert opinion on patient handover, starting to use the standard patient handover form for each patient, ensuring standardization in handover and supporting this improvement work by managers were expressed as interventions.
  Training offered; It includes the importance of patient handover, how to ensure standardization and why we should use the standard patient handover form.

SUMMARY:
This study was planned in a quasi-experimental design, focusing on the feasibility, evaluation, and implementation of patient handover between nurses, and the effect of interventions to increase their effectiveness on the patient's satisfaction with care, trust in the nurse, and the quality of nurses' patient handover.The main question it aims to answer is:

Does the intervention implemented in nurses' patient handover increase patients' satisfaction with care, its effect on their trust in nurses, and the quality of nurses' patient handover?

DETAILED DESCRIPTION:
This research was conducted between January and September 2022 at Adana City Education and Training Center.

It was carried out in the Research Hospital General Surgery Intensive Care Clinic (Intensive Care Clinic), Internal Medicine Clinic (Internal Clinic), General Surgery Clinic (Surgical Clinic). The study was carried out in a quasi-experimental design, with the control and experimental groups being the same, before the intervention, in the short term after the intervention (2 weeks after the intervention) and in the long term after the intervention (8 weeks after the intervention).

Training prepared as an expert opinion on patient handover, starting to use the standard patient handover form for each patient, ensuring standardization in handover and supporting this improvement work by managers were expressed as interventions. Training offered; It includes the importance of patient handover, how to ensure standardization and why we should use the standard patient handover form. After the training content was prepared, expert opinions were obtained from 5 people, including clinicians and academicians. The trainings were held in the meeting room of each clinic in 3 different sessions, reaching all nurses in an average of 45 minutes. The trainings were conducted interactively using written, visual and video methods. After the training, the standard patient handover form, which nurses should use in writing and verbally for each patient, was applied by the researcher at the bedside and how to use it was explained. The presentation prepared for the training was shared with nurses.

ELIGIBILITY:
Inclusion Criteria:

* Nurses using the standard patient handover form
* Nurses involved in patient handover.
* The patient over 18 years of age
* The patient understand and speak Turkish
* The patient have no hearing impairment
* The patient have no psychiatric disorder that would reduce his or her ability to comprehend and understand,
* The patient have no communication problems, have no contact isolation,
* Patients and nurses agree to participate in the research.

Exclusion Criteria:

* Nurses and patients no volunteer to participate in the research
* Nurses who do not use standard patient handover forms
* The patient under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It consists of inpatients and nurses working in the General Surgery Intensive Care Clinic, Internal Medicine Clinic and General Surgery Clinic of the training and research hospital determined between January and September 2022.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Nursing handover quality | 2 weeks and 8 weeks
  Nurses carry out written and verbal handover procedures for each patient using the standard patient handover form. Handover quality is measured by the presence of observational transferred information and the Handoff CEX Scale.

SECONDARY OUTCOMES:
Patient Trust in Nurses and Newcastle Nursing Care Satisfaction Scale Levels | 2 weeks and 8 weeks
  Evaluation of patients' Trust in Nurses and Nursing Care Satisfaction after the patient handover intervention applied to nurses. The scale is a 5-point scale consisting of 24 items including nursing care. Newcastle nursing care satisfaction scale is a 5-point scale consisting of 24 items including nursing care. It is a Likert type scale. Score evaluation is made from 0 to 100 by adding the scores of all items marked on the scale and converting them to 100. It is done based on points. A total score of 100 is considered to indicate satisfaction with all aspects of nursing care. The total score of the trust in nurses scale (minimum 5 points - maximum 30 points) is measured by summing the scores of the answers given to the questions. A high score from the scale indicates a high level of trust in nurses.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana city training and research hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gungor S, Tosun B. The Impact of Improving Clinical Patient Handover Interventions on Patient Outcomes and Handover Practices: A Complex Nursing Intervention Study. J Eval Clin Pract. 2025 Jun;31(4):e70087. doi: 10.1111/jep.70087. PMID 40323142